CLINICAL TRIAL: NCT04482543
Title: Repeated Intra-silicone Oil Injection of Methotrexate for Management of Proliferative Vitreoretinopathy Grade C; A Multi-center Study
Brief Title: Repeated Methotrexate for Proliferative Vitreoretinopathy Grade C
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shahid Beheshti University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Zahra Rabbani Khah, Head of ophthalmic research center, Shahid Beheshti University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 23454
Record Dates: First submitted 2020-07-18; First posted 2020-07-22 (Actual); Last update posted 2020-07-22 (Actual); Status verified 2020-07

CONDITIONS: Proliferative Vitreoretinopathy
MeSH Terms: conditions — Vitreoretinopathy, Proliferative | interventions — Methotrexate

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intra-silicone oil injection of 250 µg methotrexate (Active Comparator)
  Interventions: Drug: Methotrexate
- No intra-silicone oil injection of methotrexate (No Intervention)

INTERVENTIONS:
Drug: Methotrexate — Intra-silicone oil injection of 250 µg methotrexate is done at the end of surgery and is repeated at weeks 3 and 6 postoperatively.
  Arms: Intra-silicone oil injection of 250 µg methotrexate

SUMMARY:
This multicenter randomized clinical trial evaluates the effect of multiple intra-silicone oil injections of methotrexate (MTX) on rhegmatogenous retinal detachment (RRD) with grade C proliferative vitreoretinopathy (PVR).

74 eyes with the diagnosis of RRD with PVR grade C will be randomized into two groups: the intervention group and the control group. All eyes undergo pars plana vitrectomy(PPV) and intraocular injection of silicone oil (SO). At the end of the surgical procedure, intra-SO injection of 250 µg MTX will be performed in the intervention group. No intra-SO injection will be done in the control group. In the intervention group, Intra-SO injection of MTX will be repeated at 3 and 6 weeks postoperatively. Silicone oil removal will be done 3 months after surgery.Spectral-domain optical coherence tomography (SD-OCT) image of the macula will be acquired at months 3 and 6. The retinal reattachment rate at months 6 will be assessed as the main outcome measure of the study. Best corrected visual acuity, retinal reproliferation rate and adverse events are the secondary outcome measures. Comprehensive ocular examination will be performed at weeks 1, 3, 6 and at months 3, 4 and 6.

ELIGIBILITY:
Inclusion Criteria:

* Rhegmatogenous retinal detachment with proliferative vitreoretinopathy grade C

Exclusion Criteria:

* Age of under 18 years old
* Pregnancy
* Glaucoma
* Macular disorders
* Diabetic retinopathy
* Retinal vascular occlusion
* History of penetrating ocular trauma
* Giant retinal tear
* Chronic uveitis
* History of intraocular steroid injection

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 74 (Estimated)
Dates: Start 2020-08-01 (Estimated); Primary Completion 2021-07-01 (Estimated); Study Completion 2021-09-01 (Estimated)

PRIMARY OUTCOMES:
Retinal reattachment rate | 6 months
  Funduscopy

SECONDARY OUTCOMES:
Best corrected visual acuity | 6 months
  Snellen chart
Retinal reproliferation rate | 6 months
  Funduscopy
Adverse events | 6 months
  Slit-lamp, tonometry and funduscopy

CONTACTS AND LOCATIONS:
Locations (1):
- Ophthalmic Research Center, Tehran, Iran

REFERENCES:
- [Derived] Nourinia R, Safi S, Mohammadpour M, Riazi-Esfahani H, Ansari Astaneh MR, Falavarjani KG, Ramezani A, Karimi S, Fekri S, Ebrahimiadib N, Khalili Pour E, Nikkhah H, Shoeibi N, Hassanpoor N, Hosseini M, Abrishami M, Abdi F, Rahimi A, Jabbarpoor Bonyadi MH, Moradian S, Khosravi Mirzaei S, Safi H, Anvari P, Fadakar K, Mirghorbani M, Mohammadbagheri N, Hatami F, Kheiri B, Yaseri M, Khorrami Z, Ahmadieh H. Effects of repeated intra-silicone oil injections of methotrexate on proliferative vitreoretinopathy grade C: a multicenter randomized controlled trial. Sci Rep. 2024 Nov 21;14(1):28842. doi: 10.1038/s41598-024-79708-1. PMID 39572739